CLINICAL TRIAL: NCT05588063
Title: A Pilot Randomized Clinical Trial of Transcutaneous Auricular Vagus Nerve Stimulation for the Treatment of Frequently Relapsing Nephrotic Syndrome in Children
Brief Title: taVNS for FRNS in Children
Acronym: kidNEY-VNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-0488; 1R01DK131091-01A1 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-10-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Nephrotic Syndrome in Children; Minimal Change Disease; Focal Segmental Glomerulosclerosis
Keywords: vagus nerve stimulation; pediatric; nephrology
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double blinded to the investigators and participants. Unblinding will occur after all participants have completed the randomization phase of each study trial (Week 26).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intensity setting for pulse amplitude will be adjusted to the participant's tolerance (if a sensation is felt) to a maximum level of 3 on the dial indicator. The remaining settings will be stored in the device and will not need to be set for each treatment. Participants and guardians will be instructed to adjust intensity to highest level of tolerance each time the device is used and level will be logged.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation
- Sham Group (Sham Comparator): The sham device will be disabled internally so that electrical stimulation is not delivered, but the device will appear to function. Externally, the sham device will look identical to the taVNS device. The participant will be told to increase the intensity until tolerated if a sensation is felt, but will be asked to stop at a maximum level of 3. This inactive sham method was chosen because previous studies have shown that stimulation with placement of the ear clip on other parts of the ear such as the earlobe, although not innervated by the vagus nerve, results in some vagus nerve activity. Inactive sham methodology has been used in previous studies.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — The device to be used is the Roscoe Medical TENS 7000, a commercially available handheld electrical pulse generator, and an ear clip to be placed at the left ear for stimulation. Custom-made ear clips with electrode gel will be placed near the entrance to the canal of the ear to provide stimulation to the auricular branch. The handheld electrical pulse generator will be programmed to deliver electrical stimulation pulses to the cymba concha stimulating the auricular branch of the vagus nerve.
  Other Names: Roscoe TENS 7000
  Arms: Intervention Group
Device: Sham device — The device will appear to function but no electrical stimulation will be delivered.
  Other Names: Roscoe TENS 7000
  Arms: Sham Group

SUMMARY:
Children with frequently relapsing nephrotic syndrome (FRNS) are exposed to prolonged courses of steroids and other immunosuppressant medications. Given the adverse side effect profiles and variable efficacy of these medications, there is an urgent need to identify novel and safe therapies to treat nephrotic syndrome in children. Stimulation of the vagus nerve, which can be activated non invasively by transcutaneous auricular vagus nerve stimulation (taVNS), has immunomodulatory effects mediated by the inflammatory reflex and spleen. taVNS has become a therapy of interest for treating chronic immune mediated illnesses. The aims of the study are (1) To determine the feasibility of protocol implementation and tolerability of taVNS in the treatment of nephrotic syndrome in children (2) To establish proof-of-concept and generate statistical estimates of variance parameters and effect sizes for treatment response outcomes in children with nephrotic syndrome randomized to taVNS therapy compared with sham therapy (3) To investigate the effects of taVNS on inflammatory markers in children with nephrotic syndrome.

DETAILED DESCRIPTION:
Study Design A parallel, double blinded, randomized placebo controlled trial comparing daily taVNS use with sham therapy will be conducted in children 3 to17 years of age with FRNS. Thirty participants with FRNS (defined as having 2 or more relapses in 6 months within 6 months of diagnosis or 4 or more relapses in any 12 month period) will be randomized 1 to 1 to taVNS or sham therapy. Participants will be enrolled at two pediatric tertiary hospitals over a two year time period, with completion of the study by year three. All participants will perform daily taVNS therapy (active for taVNS arm or inactive for sham arm) for 5 minutes each day for a total of 26 weeks. Participants will monitor heart rate with each treatment and log home urine results. Participants will be monitored monthly with in person study visits at Weeks 8, 16 and 26 alternating with virtual remote video visits at Weeks 4, 12 and 20. Biosample specimens will be collected at baseline, 8 weeks, 16 weeks and 26 weeks. There will be a follow up period of an additional 26 weeks. All participants will be given the option to receive the active taVNS treatment at the end of the randomized period.

Intervention The device is the Roscoe Medical Transcutaneous Electrical Nerve Stimulation (TENS) 7000 unit, a FDA approved commercially available handheld electrical pulse generator. A custom-produced silicone-equivalent electrode ear clip manufactured at Feinstein will be placed at the cymba concha of the left ear with electrode gel to provide stimulation (or sham) to the auricular branch of the vagus nerve. taVNS will be performed on the left side because there is less of a risk of cardiac side effects. Maximum power density limit calculations were performed based on data from the FDA as a function of pulse width, current amplitude, electrode size, and effective impedance, suggesting an electrode size of greater than 58 mm2 must be used. The custom-made electrodes for this study are larger than this limit, thus ensuring safety. The device will be set to a frequency of 30 Hz and pulse width of 300 μs based on previous literature. All participants in both trials will perform the intervention therapy for 5 minutes each day. The timing and duration of treatment are based upon the known half-life of the biological cytokine response, previous literature demonstrating efficacy of daily 5 minute treatments and our prior work. The study period will be 26 weeks. This time period was chosen based on the definition of FRNS using a 6-month period, prior clinical trials and ethical concerns for enrolling placebo controls for a longer period of time. All participants will be told that they may or may not feel stimulation from the device. Participants will be asked not to mention any aspects of the stimulation procedures to study investigators/physicians (except to the trainer) to maintain blinding. The device has a Patient Compliance Meter that can record the number of times it was used. This will be used to monitor compliance.

taVNS Group: The intensity setting for pulse amplitude will be adjusted to the participant's tolerance (if a sensation is felt) to a maximum level of 2.5. In patients who are under the age at which they can verbalize perceptual threshold and tolerability (<5 years), the investigators will initiate intensity at the lowest setting and incrementally increase the value until the level at which perceptual threshold, defined by changes in facial expression, patient becomes fidgety, or displays behaviors which denote sensation is being perceived. Then, the intensity level will be decreased till the perceptual indicators are no longer present, and the resultant level will be used for the treatment. A maximum power density of 150 milliwatts (mW)/cm2 will be utilized for patients under the age of 5 years, a level that is substantially below the 250 mW/cm2 maximum level defined by the FDA to prevent injury. Participants and guardians will be instructed to adjust intensity to highest level of tolerance each time the device is used and level will be logged.

Sham group: The sham device will be altered internally so that electrical stimulation is not delivered, but the device will appear to function (Feinstein Bioengineering). Externally, the sham device will look identical to the taVNS device. The participant will be told to increase the intensity until tolerated if a sensation is felt, but will be asked to stop at a maximum level of 3. This inactive sham method was chosen because previous studies have shown that stimulation with placement of the ear clip on other parts of the ear such as the earlobe, although not innervated by the vagus nerve, results in some vagus nerve activity. Inactive sham methodology has been used in previous studies.

Study Phases The study will consist of three parts. Part 1 - Screening Period- up to 8 weeks. Informed consent/assent will be obtained at screening prior to the conduct of any study-related procedures. Participants will be screened to confirm inclusion/exclusion criteria are met. Participants must be off steroid treatment for 14 days prior to Day 1 and the participant must be in remission (negative urine protein creatinine (UPC) on first morning urine) on Day 1.

Part 2 - Randomized Control Period - 26 weeks: Thirty participants with FRNS who meet all of the eligibility criteria will be randomized 1:1 to either taVNS or sham treatment. A trainer will instruct the parent/guardian on use of the device at the randomization visit. Participants will use the intervention device as directed for 5 minutes per day for 26 weeks. Participants will be monitored monthly with in-person study visits at Weeks 8, 16 and 26 alternating with virtual remote video visits at Weeks 4, 12 and 20. The visit window will be +/- 7 days. At each in person visit, the following will be conducted:

* Vital signs and physical examination
* Assessment for nephrotic syndrome relapses. Home urine protein logs will be reviewed.
* Blood and urine samples will be collected at each in person visit.
* Assessment of study intervention adherence. Parents/guardians will meet with the trainer and will be reoriented on taVNS device use at each visit as a safety measure. The device counter number will be recorded as a measure of adherence.
* Monitor for adverse events and tolerability: Parents/guardians will share a study log with investigators, which describes daily taVNS use, side effects, and any changes in heart rate.

At each virtual remote video visit, we will observe the participant while doing the intervention procedure, assess for nephrotic syndrome relapses, and monitor for any adverse events.

There will be a 4 week acclimation phase. If the participant relapses during this period, they will be treated with standard of care steroids and continue the intervention. If the participant relapses a second time or relapses after the acclimation phase, they will be terminated from the randomization phase and entered into the follow up period.

Part 3 - Follow Up Period - 26 weeks: At the completion of the randomized period, participants will be followed for an additional 26 weeks to assess clinical status. For those who stop the intervention, study visits will occur in-person during regularly scheduled clinical visits or via telehealth visit every 8 weeks, whichever is sooner. Participants will be assessed for the number of nephrotic syndrome relapses and home urine protein logs will be reviewed. First morning UPC will be recorded. All participants will be given the option to receive the active taVNS treatment at the end of the randomized period. Unblinding of treatment assignment from the randomized phase will not occur prior to consent for open-label use. As open-label extension trials may introduce significant bias, data obtained from these participants will not be considered part of this research and no statistical analysis will be carried out. However, clinical status and safety will continue to be monitored. In person study visits will occur every 8 weeks for those continuing use of taVNS.

Participant Discontinuation/Withdrawal from the Study Participation is completely voluntary and participants may decide to withdraw at any time. If a participant becomes steroid dependent at any point, they will be withdrawn from the study by investigators and offered alternative immunosuppressive therapy as per standard of care. If a participant in the SRNS group has deterioration in clinical status (e.g. worsening edema, rising creatinine), the treating physician may recommend withdrawal from the study at any point.

The pilot trial is not powered to determine statistically significant differences in efficacy endpoints comparing taVNS with sham therapy. Efficacy analyses will be reserved for the subsequent main trial. Rather, sample sizes were chosen to appropriately assess the feasibility, tolerability and variance effect size endpoints of the pilot trials.

ELIGIBILITY:
Inclusion Criteria:

* FRNS
* Age 3-17 years
* Glomerular filtration rate (eGFR) ≥30 ml/min/1.73 m2
* Minimal change disease (MCD) or focal segmental glomerulosclerosis (FSGS) diagnosis (clinical diagnosis or per biopsy)
* Steroid sensitive nephrotic syndrome (prior history of remission within 4 weeks of steroid therapy)
* In remission at time of enrollment (remission defined as UPC <0.2 or negative dipstick for 3 consecutive days)
* Informed consent from the parent or guardian and assent from a minor of ≥ 7. years

Exclusion Criteria:

* Secondary forms of nephrotic syndrome
* SRNS
* Steroid dependent nephrotic syndrome (relapse within 14 days of stopping steroids or relapse while on steroids)
* Exposure to steroids within 14 days of enrollment
* Receiving any standing immunosuppression (previous exposure > 2 months allowed and/or B cell repletion)
* Any known inflammatory condition (e.g. systemic lupus erythematosis)
* History of cardiac disease (arrhythmias, structural/functional abnormalities)
* Implantable electronic devices
* Pregnancy
* Participants/guardians or participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Success of Pilot Trial | Baseline through 26 weeks
  1. Unsuccessful, main study not practicable (1) None of the benchmarks are met, or (2) One or more of the benchmarks are not met and there is low likelihood of reaching benchmarks even with protocol modifications or (3) Serious adverse events related to the treatment.
  2. Probable Success main study practicable with modifications to protocol. One or more of the benchmarks are not met, but there is a high likelihood that the benchmark can be met with protocol modifications.
  3. Successful main study practicable without modifications. All of the benchmarks are met.

SECONDARY OUTCOMES:
Proof-of-Concept Decision Criteria using relative risk for relapse | Baseline through 26 weeks
  The decision to move forward with a larger trial will be made based on pre-determined proof of concept decision criteria. Once data from the pilot trial is observed and collected, 1,000 bootstrap resamples with replacement will be carried out to construct the empirical 95% confidence interval (CI) for the relative risk. Using a non-parametric approach, the lower 2.5th percentile and upper 97.5th percentile will be used to construct the CI, and a GO or NO GO decision to conduct the larger scale trial will be made based on a primary end point. The primary end-point is no relapses within 26 weeks. Based on previous literature, it is presumed that 50% in the intervention arm and 25% of those in sham therapy will reach the primary end-point in each trial, which is equivalent to a relative risk of 2.0.
Estimates of Variance for proportion with nephrotic syndrome relapse | Baseline through 26 weeks
  Frequency counts and proportions with 95 percent confidence intervals
Estimates of Variance for time to nephrotic syndrome relapse | Baseline through 26 weeks
  Mean and standard deviation
Estimates of Variance for time to achieve remission once a relapse occurs | Baseline through 26 weeks
  Mean and standard deviation
Recruitment rate | Baseline through 26 weeks
  Percent
Drop out rate | Baseline through 26 weeks
  Percent
Rate of completion of study | Baseline through 26 weeks
  Percent
Successful double-blinding | Baseline through 26 weeks
  Percent
Treatment adherence from home logs | Baseline through 26 weeks
  Percent
Adverse events | Baseline through 26 weeks
  Percent
Incidence of withdrawal due to adverse events | Baseline through 26 weeks
  Percent
Cytokines | Baseline through 26 weeks
  Tumor necrosis factor (TNF), interleukin (IL)-6 mean and standard deviation
Anti-nephrin antibodies | Baseline through 26 weeks
  Mean and standard deviation
Whole monocyte stimulation assay | 0 hour and 2 hours
  Intracellular cytokines at 0 and 2 hours

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Informed consent documents for the clinical trials will be available on clinical trials.gov. Data will be available from the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study closure